CLINICAL TRIAL: NCT05041608
Title: Endoscopic Surgery for Gastrointestinal Disorders: A Multicenter Registry Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Advanced Endoscopy Research, Robert Wood Johnson Medical School Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2020002798
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Achalasia; Gastric Outlet Obstruction; Gastroparesis; GERD; Reflux; Fistula; Benign Neoplasm
Keywords: POEM; ESD; STER; EFTR; EMR; NOTES; TIF; Capsule Endoscopy; Endoscopic suturing; Endoscopic Fistula Closure; ZPOEM; GPOEM
MeSH Terms: conditions — Esophageal Achalasia; Gastric Outlet Obstruction; Gastroparesis; Gastroesophageal Reflux; Fistula; Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects undergoing Endoscopic Surgery: These procedures include: POEM (Peroral Endoscopic Myotomy) for Achalasia, G-POEM (Gastric Peroral Endoscopic Myotomy) for gastric outlet obstruction, Z-POEM (Peroral endoscopic myotomy for Zenker's Diverticulum), EMR (Endoscopic Mucosal Resection), ESD (Endoscopic submucosal dissection), STER (Submucosal tunneling endoscopic resection), NOTES (Natural Orifice Translumenal Endoscopic Surgery), TIF (Transoral Incisionless Fundoplication), Endoscopic Fistula Closure, Endoscopic Suturing, Capsule Endoscopy and EFTR (Endoscopic full-thickness resection).
  Interventions: Procedure: Endoscopic Surgery

INTERVENTIONS:
Procedure: Endoscopic Surgery — These procedures include: POEM (Peroral Endoscopic Myotomy) for Achalasia, G-POEM (Gastric Peroral Endoscopic Myotomy) for gastric outlet obstruction, Z-POEM (Peroral endoscopic myotomy for Zenker's Diverticulum), EMR (Endoscopic Mucosal Resection), ESD (Endoscopic submucosal dissection), STER (Submucosal tunneling endoscopic resection), NOTES (Natural Orifice Translumenal Endoscopic Surgery), TIF (Transoral Incisionless Fundoplication), Endoscopic Fistula Closure, Endoscopic Suturing, Capsule Endoscopy and EFTR (Endoscopic full-thickness resection).

SUMMARY:
Currently, there is limited multi-center data on endoscopic surgery outcomes in western populations.

Evaluation of these measurement would help the investigators compare them to conventional treatment modalities within current tertiary facilities; and consequently help the investigators identify appropriate treatment techniques and improve clinical management of patients at Rutgers RWJMS.

The purpose of this retrospective registry study is to assess long term data on efficacy, safety and clinical outcome of Endoscopic Surgery within the gastrointestinal tract.

DETAILED DESCRIPTION:
Our tertiary-care institution performs clinically-indicated various Endoscopic Surgery procedures gastrointestinal indications in more than 800-1000 patients annually.

The study investigators would collect data on a large sample size of subjects undergoing various endoscopic resection procedures such as POEM (Peroral Endoscopic Myotomy), EMR (Endoscopic Mucosal Resection), ESD (Endoscopic submucosal dissection), STER (Submucosal tunneling endoscopic resection), NOTES (Natural Orifice Translumenal Endoscopic Surgery), TIF (Transoral Incisionless Fundoplication), Endoscopic Fistula Closure, Endoscopic Suturing, Capsule Endoscopy and EFTR (Endoscopic full-thickness resection). Clinical metrics will be collected including procedure times, length of follow-up, specific tumor characteristics, resection method, pathology results, procedural complications, additional therapy required, and disease-free survival time.

Various endoscopic surgical procedures are less invasive than traditional surgery, have fewer side effects and provide better efficacy. Moreover, they can be available to patients who are ineligible for surgery or who have refused more aggressive surgical intervention.

They improve quality of life and extend survival duration.

Endoscopic surgery procedures can be an appropriate approach in many gastrointestinal disorders including early neoplasms, challenging adenomas or sub-epithelial lesions that requires the resection of the superficial layers, mucosa and submucosa, or full thickness resection of the tract wall.

Currently, there is limited multi-center data on endoscopic surgery outcomes in western populations.

Evaluation of these measurement would help the investigators compare them to conventional treatment modalities within current tertiary facilities; and consequently help the investigators identify appropriate treatment techniques and improve clinical management of patients at Rutgers RWJMS.

The purpose of this retrospective registry study is to assess long term data on efficacy, safety and clinical outcome of Endoscopic Surgery within the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing Endoscopic Surgery

Exclusion Criteria:

* Subjects not undergoing Endoscopic Surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing Endoscopic Surgery for various Gastrointestinal indications
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Efficacy of procedure | Upto 1 year
  Technical and clinical success rate
Safety of procedure | Upto 1 year
  Type, frequency and intensity of adverse events

SECONDARY OUTCOMES:
Quality of Life after procedure | Upto 1 year
  Chart Review of quality-of-life improvement and overall survival duration

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Advanced Endoscopy Research, Robert Wood Johnson Medical School Rutgers University
Locations (1):
- Advanced Endoscopy Research, Robert Wood Johnson Medical School Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers.

REFERENCES:
- [Derived] Shahid HM, Bareket R, Tyberg A, Sarkar A, Simon A, Gurram K, Gress FG, Bhenswala P, Chalikonda D, Loren DE, Kowalski TE, Kumar A, Vareedayah AA, Abhyankar PR, Parker K, Gabr MM, Nieto J, De Latour R, Zolotarevsky M 5th, Barber J, Zolotarevsky E, Vazquez-Sequeiros E, Gaidhane M, Andalib I, Kahaleh M. Comparing the Safety and Efficacy of Two Commercially Available Single-Use Duodenoscopes: A Multicenter Study. J Clin Gastroenterol. 2023 Sep 1;57(8):798-803. doi: 10.1097/MCG.0000000000001752. PMID 35997700
- [Derived] Shah-Khan SM, Zhao E, Tyberg A, Sarkar S, Shahid HM, Duarte-Chavez R, Gaidhane M, Kahaleh M. Endoscopic Ultrasound-Directed Transgastric ERCP (EDGE) Utilization of Trends Among Interventional Endoscopists. Dig Dis Sci. 2023 Apr;68(4):1167-1177. doi: 10.1007/s10620-022-07650-1. Epub 2022 Aug 10. PMID 35947304